CLINICAL TRIAL: NCT00780754
Title: Effect of 5α Reductase Inhibitor Dutasteride on the Prevention of the Prostate Cancer in Men With High Grade Intraepithelial Neoplasia of the Prostate
Brief Title: Prevention of Prostate Cancer With Dutasteride in Case of High Grade PIN Neoplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaunas University of Medicine (Other)
Responsible Party: Principal Investigator, Stasys Auskalnis, doctor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BE-2-27
Record Dates: First submitted 2008-10-26; First posted 2008-10-28 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2008-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; chemoprevention; dutasteride
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dutasteride (Experimental): treatment group
  Interventions: Drug: dutasteride; Procedure: prostate biopsy
- watchful waiting strategy (Active Comparator)
  Interventions: Procedure: prostate biopsy

INTERVENTIONS:
Drug: dutasteride — 0.5mg
  Arms: dutasteride
Procedure: prostate biopsy — prostate biopsy

SUMMARY:
Patients with diagnosis of HPIN were enrolled. Patients were randomized into two groups: dutasteride treatment group and watchful waiting strategy group. According to the study protocol the subjects would undergo 10 core biopsies after 6, 12, 24, and 36 months after randomization.

There are assessed the rate of prostate cancer at repeated transrectal ultrasound guided biopsies and the effect of 5 alfa reductase inhibitor (dutasteride) on prevention of prostate cancer development for patients with high grade intraepithelial neoplasia (HPIN).

ELIGIBILITY:
Inclusion Criteria:

1. Age - 40-80 years
2. HPIN on prostate biopsy specimens
3. PSA below 20ng/ml
4. No hormone therapy or radiation in pelvic region
5. No previous treatment with 5alfa reductase inhibitors
6. Signed Subject Information and Informed Subject Consent Form.

Exclusion Criteria:

1. Not compensate cardiovascular, pulmonary, hepatic or renal functions, neurological, psychiatric disease, sepsis, etc.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
rate of prostate cancer at repeated transrectal ultrasound guided biopsies in case of HPIN | 6, 12, 24, and 36 months

SECONDARY OUTCOMES:
effect of 5 alfa reductase inhibitor (dutasteride) on prevention of prostate cancer development for patients with high grade intraepithelial neoplasia (HPIN). | 6, 12, 24, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Daimantas Milonas, assist professor, Principal Investigator — Kaunas Medical University
Locations (1):
- Urology dep. of Kaunas University of Medicine, Kaunas, Lithuania